CLINICAL TRIAL: NCT06058247
Title: Reducing In-Hospital and 60-Day Mortality in Critically Ill Patients After Surgery With Strict Nutritional Supplementation: A Prospective, Single-Labeled, Randomized Controlled Trial
Brief Title: Reducing In-Hospital and 60-Day Mortality in ICU Patients After Surgery With Strict Nutritional Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Eun Young Kim, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUMIS_02
Record Dates: First submitted 2023-09-05; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Protein-Energy Malnutrition
MeSH Terms: conditions — Protein-Energy Malnutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active nutritional supplementation (Experimental): The participants in active nutritional supplementation arm received nutritional support targeting specific protein (over 1.5 g/kg/day) and calorie intake (over 20 kcal/kg/day), with consultation from the nutritional support team and the initiation of nutritional supplementation on the same day as intensive care unit admission.
  Interventions: Dietary Supplement: Active nutritional supplementation
- Conventional nutritional supplementation (Experimental): The participants in conventional nutritional supplementation arm underwent conventional nutrition management without specific protein or caloric targets.
  Interventions: Dietary Supplement: Conventional nutritional supplementation

INTERVENTIONS:
Dietary Supplement: Active nutritional supplementation — The participants in active nutritional supplementation arm received consultation from the nutritional support team (NST) upon ICU admission, and nutritional supplementation was initiated on the same day.
  NST is a multidisciplinary support team comprised of physicians, nurses, dietitians, and pharmacists, which assesses the nutritional status of patients, and provides recommendations for nutritional therapy. Targets in the participants in active nutritional supplementation arm were protein supplementation at over 1.5 g/kg/day, calorie provision at over 20 kcal/kg/day, and energy adequacy of at least 80%. Energy target was estimated by multiplying the resting energy expenditure using the Harris and Benedict equation by an activity factor of 1.3 and a stress factor of 1.1. Actual body weight was used as the body weight for patients with a percent of ideal body weight (PIBW) of less than 120%, while adjusted body weight was used for patients with a PIBW greater than or equal to 120%.
  Arms: Active nutritional supplementation
Dietary Supplement: Conventional nutritional supplementation — The participants in conventional nutritional supplementation arm received conservative nutritional management without specific protein or caloric targets.
  Arms: Conventional nutritional supplementation

SUMMARY:
Malnutrition in critically ill patients is a global concern due to its association with increased infectious complications, prolonged hospital stays, and higher morbidity rates. Patients who undergo abdominal surgery are particularly vulnerable due to alterations in gastrointestinal function and prolonged fasting. Despite the significance of proper nutrition, guidelines remain broad, and practical implementation is often inadequate.

The investigators aimed to assess the effects of strict nutritional provision, targeting an energy adequacy of 80% or more and a protein intake of at least 1.5 g/kg/day, on in-hospital and 60-day mortality.

DETAILED DESCRIPTION:
During the acute phase of critical illness, patients experience metabolic and physiological changes that affects their nutrition status. One prominent feature is the activation of stress hormones and inflammatory mediators, which contribute to a negative nitrogen balance, increased gluconeogenesis, and accelerated muscle proteolysis. Among these patients, those who undergo abdominal surgery are particularly vulnerable to malnutrition as they experience alterations in the structural barrier of the gastrointestinal tract, impaired nutrient absorption, and prolonged fasting due to concerns such as the integrity of an anastomosis. Thus, appropriate nutritional therapy should be prioritized for critically ill patients following abdominal surgery, and it should include adequate nutritional support to preserve lean body mass and organ function.

Despite the importance of nutritional supply, the recommendations for protein or calorie intake vary according to different guidelines, and this is the same for surgical patients. Additionally, some patients experience a delay in initiating nutritional support, and several studies reported that only 39 - 63% of the intended energy and 45 - 55% of the prescribed protein are being administered to critically ill patients during the acute phase. Furthermore, recent randomized controlled trials reported conflicting results with current guidelines, with some suggesting that lower calorie or higher protein dose administrations did not significantly impact clinical outcomes and may even worsen the outcomes for certain patient groups. Thus, the optimal nutritional provision target during the acute phase of critical illness, particularly for surgical patients, remains controversial, and there is no standardized protocol.

In our previous study, the malnutrition status upon admission, indicated by a modified Nutrition Risk in the Critically Ill (mNUTRIC) score of 5 or higher, and low energy adequacy during intensive care unit (ICU) stay were identified as mortality predictors in critically ill patients following abdominal surgery. The investigators aimed to assess the effects of strict nutritional provision, targeting an energy adequacy of 80% or more and a protein intake of at least 1.5 g/kg/day, on in-hospital and 60-day mortality. Additionally, the investigators investigated the appropriate target for nutrition support in critically ill patients who undergo abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted after abdominal surgery to our institution's surgical ICU
* They were enrolled regardless of the surgical method, either open, laparoscopy, or robotic.

Exclusion Criteria:

* aged under 18 years
* underwent surgery under local or regional anesthesia
* pregnant
* readmitted to the ICU
* diagnosed with renal failure and receiving renal replacement therapy
* lacked individual data necessary to calculate the mNUTRIC score measured at ICU admission
* failed to provide informed consent, or with 'do-not-resuscitate' status.
* the patient was discharged or expired within 48 hours of ICU admission
* patients diagnosed with multiorgan failure, represented by a high Sequential Organ Failure Assessment (SOFA) score (≥9) upon ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
60-day mortality rate | Participants were followed upto 60th day after surgery
  Proportion of patients who died within 60 days after surgery among participants

SECONDARY OUTCOMES:
In-hospital mortality rate | Participants were followed upto 60th day after surgery
  Proportion of patients who died during the hospitalization period
Incidence of postoperative complications | Participants were followed upto 60th day after surgery
  Proportion of patients who died within 60 days after surgery among participants

CONTACTS AND LOCATIONS:
Overall Officials: Hye sung Kim, Study Director — The Catholic University of Korea
Locations (1):
- Division of Trauma and Surgical Critical Care, Department of Surgery, Seoul St. Mary's Hospital, Seoul, Seocho-gu, Banpo-dong Banpodaero 222, South Korea